CLINICAL TRIAL: NCT01565941
Title: Heart And Lung Failure - Pediatric INsulin Titration Trial (HALF-PINT)
Brief Title: Heart And Lung Failure - Pediatric INsulin Titration Trial
Acronym: HALF-PINT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Agus, Associate Professor of Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00002310; U01HL107681 (NIH)
Record Dates: First submitted 2012-03-21; First posted 2012-03-29 (Estimated); Results first posted 2017-12-11 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Respiratory Failure
Keywords: Cardiovascular; Respiratory; Failure; Heart; Lung; Continuous glucose monitoring; Tight glycemic control; Subcutaneous; Insulin; Algorithm
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tight Glycemic Control 1 (TGC-1) (Active Comparator): Approximately half of the subjects randomized into HALF-PINT will be randomized into TGC-1 which will seek to maintain the subject's blood sugar between 80-110 mg/dL. Intravenous insulin may be administered per insulin algorithm.
  Interventions: Drug: Insulin
- Tight Glycemic Control 2 (TGC-2) (Active Comparator): Approximately half of the subjects randomized into HALF-PINT will be randomized into TGC-2 which will seek to maintain the subject's blood sugar between 150-180 mg/dL. Intravenous insulin may be administered per insulin algorithm.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — IV insulin titration to target a blood glucose of 80-110 mg/dL
  Arms: Tight Glycemic Control 1 (TGC-1)
Drug: Insulin — IV insulin titration to target a blood glucose of 150-180 mg/dL
  Arms: Tight Glycemic Control 2 (TGC-2)

SUMMARY:
Stress hyperglycemia, a state of abnormal metabolism with supra-normal blood glucose levels, is often seen in critically ill patients. Tight glycemic control (TGC) was originally shown to reduce morbidity and mortality in a landmark randomized clinical trial (RCT) of adult critically ill surgical patients but has since come under intense scrutiny due to conflicting results in recent adult trials. One pediatric RCT has been published to date that demonstrated survival benefit but was complicated by an unacceptably high rate of severe hypoglycemia. The Heart And Lung Failure - Pediatric INsulin Titration (HALF-PINT) trial is a multi-center, randomized clinical treatment trial comparing two ranges of glucose control in hyperglycemic critically ill children with heart and/or lung failure. Both target ranges of glucose control fall within the range of "usual care" for critically ill children managed in pediatric intensive care units.

The purpose of the study is to determine the comparative effectiveness of tight glycemic control to a target range of 80-110 mg/dL (TGC-1, 4.4-6.1 mmol/L) vs. a target range of 150-180 mg/dL (TGC-2, 8.3-10.0 mmol/L) on hospital mortality and intensive care unit (ICU) length of stay (LOS) in hyperglycemic critically ill children with cardiovascular and/or respiratory failure. This will be accomplished using an explicit insulin titration algorithm and continuous glucose monitoring to safely achieve these glucose targets. Both groups will receive identical standardized intravenous glucose at an age-appropriate rate in order to provide basal calories and mitigate hypoglycemia. Insulin infusions will be titrated with an explicit algorithm combined with continuous glucose monitoring using a protocol that has been safely implemented in 490 critically ill infants and children.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular failure and/or respiratory failure:

  1. Cardiovascular Failure: Dopamine or dobutamine > 5 mcg/kg/min, or any dose of epinephrine, norepinephrine, phenylephrine, milrinone or vasopressin if used to treat hypotension.
  2. Respiratory Failure: Acute mechanical ventilation via endotracheal tube or tracheostomy.
* Age >= 2 weeks and corrected gestational age >= 42 weeks
* Age < 18 years (has not yet had 18th birthday)

Exclusion Criteria:

* No longer has cardiovascular or respiratory failure (as defined in inclusion criterion 1), or is expected to be extubated in the next 24 hours
* Expected to remain in ICU < 24 hours
* Previously randomized in HALF-PINT
* Enrolled in a competing clinical trial
* Family/team decision to limit/redirect from aggressive ICU technological support
* Chronic ventilator dependence prior to ICU admission (non-invasive ventilation and ventilation via tracheostomy overnight or during sleep are acceptable)
* Type 1 or 2 diabetes
* Cardiac surgery within prior 2 months or during/planned for this hospitalization (extra-corporeal life support or non-cardiac surgery is acceptable)
* Diffuse skin disease that does not allow securement of a subcutaneous sensor
* Therapeutic plan to remain intubated for >28 days
* Receiving therapeutic cooling with targeted body temperatures <34 degrees Celsius
* Current or planned ketogenic diet
* Ward of the state
* Pregnancy

Ages: 2 Weeks to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 713 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael SD Agus, MD, Principal Investigator — Boston Children's Hospital; Vinay M Nadkarni, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (35):
- United States (33):
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Children's Hospital of Los Angelos, Los Angeles, California
  - Mattel Children's Hospital, Los Angeles, California
  - Children's Hospital & Research Center of Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Nemours/A.I DuPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital pf Chicago, Chicago, Illinois
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - North Shore LIJ Cohen Children's Medical Center, New Hyde Park, New York
  - Morgan Stanley Children's Hospital of New York, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke Children's Hospital and Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical City Children's Dallas, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Royal Children's Hospital, Melbourne, Victoria, Australia
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agus MS, Hirshberg E, Srinivasan V, Faustino EV, Luckett PM, Curley MA, Alexander J, Asaro LA, Coughlin-Wells K, Duva D, French J, Hasbani N, Sisko MT, Soto-Rivera CL, Steil G, Wypij D, Nadkarni VM. Design and rationale of Heart and Lung Failure - Pediatric INsulin Titration Trial (HALF-PINT): A randomized clinical trial of tight glycemic control in hyperglycemic critically ill children. Contemp Clin Trials. 2017 Feb;53:178-187. doi: 10.1016/j.cct.2016.12.023. Epub 2016 Dec 30. PMID 28042054
- [Derived] LaRovere KL, Asaro LA, Coughlin-Wells K, Nadkarni VM, Agus MSD; Heart and Lung Failure-Pediatric Insulin Titration (HALF-PINT) Study Investigators. Blood Glucose Range for Hyperglycemic PICU Children With Primary Neurologic Diagnoses: Analysis of the Heart and Lung Failure-Pediatric Insulin Titration (HALF-PINT) Trial. Pediatr Crit Care Med. 2025 Apr 1;26(4):e432-e446. doi: 10.1097/PCC.0000000000003689. Epub 2025 Feb 5. PMID 39907523
- [Derived] Yang JO, Zinter MS, Pellegrini M, Wong MY, Gala K, Markovic D, Nadel B, Peng K, Do N, Mangul S, Nadkarni VM, Karlsberg A, Deshpande D, Butte MJ, Asaro L, Agus M, Sapru A; Study Site Investigators for CAF-PINT. Whole blood transcriptomics identifies subclasses of pediatric septic shock. Crit Care. 2023 Dec 8;27(1):486. doi: 10.1186/s13054-023-04689-y. PMID 38066613
- [Derived] Yang JO, Zinter MS, Pellegrini M, Wong MY, Gala K, Markovic D, Nadel B, Peng K, Do N, Mangul S, Nadkarni VM, Karlsberg A, Deshpande D, Butte MJ, Asaro L, Agus M, Sapru A. Whole Blood Transcriptomics Identifies Subclasses of Pediatric Septic Shock. Res Sq [Preprint]. 2023 Aug 28:rs.3.rs-3267057. doi: 10.21203/rs.3.rs-3267057/v1. PMID 37693502
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Zinter MS, Markovic D, Asaro LA, Nadkarni VM, McQuillen PS, Sinha P, Matthay MA, Jeschke MG, Agus MSD, Sapru A; CAF-PINT Investigators of the PALISI Network. Tight Glycemic Control, Inflammation, and the ICU: Evidence for Heterogeneous Treatment Effects in Two Randomized Controlled Trials. Am J Respir Crit Care Med. 2023 Apr 1;207(7):945-949. doi: 10.1164/rccm.202210-1988LE. No abstract available. PMID 36656551
- [Derived] Hirshberg EL, Alexander JL, Asaro LA, Coughlin-Wells K, Steil GM, Spear D, Stone C, Nadkarni VM, Agus MSD; HALF-PINT Study Investigators. Performance of an Electronic Decision Support System as a Therapeutic Intervention During a Multicenter PICU Clinical Trial: Heart and Lung Failure-Pediatric Insulin Titration Trial (HALF-PINT). Chest. 2021 Sep;160(3):919-928. doi: 10.1016/j.chest.2021.04.049. Epub 2021 Apr 29. PMID 33932465
- [Derived] LaMarra D, French J, Bailey C, Sisko MT, Coughlin-Wells K, Agus MSD, Srinivasan V, Nadkarni VM; Heart And Lung Failure-Pediatric INsulin Titration (HALF-PINT) Study Investigators. A Novel Framework Using Remote Telesimulation With Standardized Parents to Improve Research Staff Preparedness for Informed Consent in Pediatric Critical Care Research. Pediatr Crit Care Med. 2020 Dec;21(12):e1042-e1051. doi: 10.1097/PCC.0000000000002484. PMID 32740181
- [Derived] Biagas KV, Hinton VJ, Hasbani NR, Luckett PM, Wypij D, Nadkarni VM, Agus MSD; HALF-PINT trial study investigators; PALISI Network. Long-Term Neurobehavioral and Quality of Life Outcomes of Critically Ill Children after Glycemic Control. J Pediatr. 2020 Mar;218:57-63.e5. doi: 10.1016/j.jpeds.2019.10.055. Epub 2020 Jan 3. PMID 31910992
- [Derived] Srinivasan V, Hasbani NR, Mehta NM, Irving SY, Kandil SB, Allen HC, Typpo KV, Cvijanovich NZ, Faustino EVS, Wypij D, Agus MSD, Nadkarni VM; Heart and Lung Failure-Pediatric Insulin Titration (HALF-PINT) Study Investigators. Early Enteral Nutrition Is Associated With Improved Clinical Outcomes in Critically Ill Children: A Secondary Analysis of Nutrition Support in the Heart and Lung Failure-Pediatric Insulin Titration Trial. Pediatr Crit Care Med. 2020 Mar;21(3):213-221. doi: 10.1097/PCC.0000000000002135. PMID 31577692
- [Derived] Agus MS, Wypij D, Hirshberg EL, Srinivasan V, Faustino EV, Luckett PM, Alexander JL, Asaro LA, Curley MA, Steil GM, Nadkarni VM; HALF-PINT Study Investigators and the PALISI Network. Tight Glycemic Control in Critically Ill Children. N Engl J Med. 2017 Feb 23;376(8):729-741. doi: 10.1056/NEJMoa1612348. Epub 2017 Jan 24. PMID 28118549

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Started | 360 | 353
Completed | 349 | 349
Not Completed | 11 | 4
Not completed — Withdrawn by parent/guardian | 3 | 2
Not completed — Randomized; did not receive intevention | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2) | Total
Number analyzed (Participants) | 349 | 349 | 698
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 349 | 349 | 698
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 5.5 [1.4 to 12.5] | 6.7 [1.7 to 12.8] | 6.2 [1.6 to 12.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 169 | 333
  Male | 185 | 180 | 365
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2
  United States | 348 | 348 | 696

OUTCOME MEASURES:

1. Primary Outcome: ICU-Free Days
Description: 28-day hospital mortality-adjusted ICU length of stay.
Time Frame: Study day 28
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Days | 20 [1.0 to 24.2] | 19.4 [7.1 to 23.9]

2. Secondary Outcome: 90-day Hospital Mortality
Description: In order to enable direct comparisons between data gathered in HALF-PINT and the prior adult NICE-SUGAR trial, we will collect data on 90-day hospital mortality.
Time Frame: 90 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 52 | 40

3. Secondary Outcome: 28-day Hospital Mortality
Description: We will collect data on 28-day hospital mortality.
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 47 | 32

4. Secondary Outcome: Accumulation of Multiple Organ Dysfunction Syndrome (MODS)
Description: Accumulation of MODS during the 28 days following randomization will be measured. MODS is defined as the concurrent dysfunction of two or more organ systems (e.g., acute lung injury and renal failure). The clinical relevance of MODS as a surrogate outcome measure is well recognized in the intensive care community, and there is a clear relationship between the number of dysfunctional organ systems and the risk of death in critically ill children.
Time Frame: 28 days after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 326 | 324

5. Secondary Outcome: Ventilator-Free Days
Description: Ventilator-free days during the 28 days following randomization encompasses both reduction in the duration of ventilation and improvement in mortality. The end of the subject's duration of ventilation is defined as the date/time of extubation for subjects who are intubated, or the date/time of the discontinuation of mechanical ventilation for subjects with tracheostomy.
Time Frame: 28 days following randomization
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Days | 21.8 [8.4 to 25.0] | 20.9 [11.9 to 24.4]

6. Secondary Outcome: Developmental Neurobehavioral Outcomes: VABS-II Composite
Description: Reliable, reproducible measures of adaptive functioning, behavior and quality of life will be used to determine outcomes at baseline (CBCL, PedsQL) and at one year after ICU discharge (Vineland-II, CBCL, PedsQL). The goal of baseline data collection is to assess pre-ICU health and quality of life. The results of the Vineland Adaptive Behavior Scales, Second Edition (VABS-II) are reported. Scores range from 20-160, with higher scores being better.
Time Frame: One year after ICU course
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 97 | 111
Score on a scale | 79.9 (25.5) | 79.4 (26.9)

7. Secondary Outcome: Participants With Device-Related or Non-Device Related Nosocomial Infection
Description: We will use Centers for Disease Control's (CDC) most recently published definitions for the following nosocomial infections attributable to the ICU stay: total bloodstream infections including Central Venous Line (CVL)-associated bloodstream infections (BSI), respiratory tract infections including ventilator-associated pneumonias, urinary tract infections, and wound infections that occur in the ICU or within 48 hours of discharge to the non-ICU inpatient unit.
Time Frame: Up to 48 hours after ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 12 | 4

8. Secondary Outcome: Incidence of Catheter-Associated Bloodstream Infection
Description: We will use Centers for Disease Control's (CDC) most recently published definition for the following nosocomial infection attributable to the ICU stay: Central Venous Line (CVL)-associated bloodstream infections (BSI) that occur in the ICU or within 48 hours of discharge to the non-ICU inpatient unit. This device-related infection will be counted per 1,000 device days.
Time Frame: Up to 48 hours after ICU discharge
Measure: Number; unit: Infections/1000 CVC days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Infections/1000 CVC days | 1.94 | 0

9. Secondary Outcome: Incidence of Catheter-Associated Urinary Tract Infection
Description: We will use Centers for Disease Control's (CDC) most recently published definition for the following nosocomial infection attributable to the ICU stay: urinary tract infections that occur in the ICU or within 48 hours of discharge to the non-ICU inpatient unit. This device-related infection will be counted per 1,000 device days.
Time Frame: Up to 48 hours after ICU discharge
Measure: Number; unit: Infections/1000 bladder catheter days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Infections/1000 bladder catheter days | 2.19 | 1.79

10. Secondary Outcome: Incidence of Ventilator-Associated Pneumonia
Description: We will use Centers for Disease Control's (CDC) most recently published definition for the following nosocomial infection attributable to the ICU stay: respiratory tract infections including ventilator-associated pneumonias that occur in the ICU or within 48 hours of discharge to the non-ICU inpatient unit. This device-related infection will be counted per 1,000 device days.
Time Frame: Up to 48 hours after ICU discharge
Measure: Number; unit: Infections/1000 ventilator days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Infections/1000 ventilator days | 0.94 | 0

11. Secondary Outcome: Incidence of Wound Infection Incidence of Wound Infection
Description: We will use Centers for Disease Control's (CDC) most recently published definition for the following nosocomial infection attributable to the ICU stay: wound infections that occur in the ICU or within 48 hours of discharge to the non-ICU inpatient unit. This non-device-related infection will be counted per 1,000 ICU days.
Time Frame: Up to 48 hours after ICU discharge
Measure: Number; unit: Infections/1000 ICU days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Infections/1000 ICU days | 0 | 0

12. Secondary Outcome: Participants With Severe Hypoglycemia (<40 mg/dL), Unrelated to Insulin Infusion (Insulin Algorithm Safety)
Description: Hypoglycemia will be tracked and reported according to three ranges: severe (<40 mg/dL), moderate (40-49 mg/dL) and mild (50-59 mg/dL). As insulin infusion can cause slight changes to serum potassium concentration, hypokalemia <2.5 mmol/L will also be tracked.
Time Frame: Participants will be followed for the duration of ICU stay, an expected average of 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 5 | 6

13. Secondary Outcome: Participants With Severe Hypoglycemia (<40 mg/dL), Related to Insulin Infusion (Insulin Algorithm Safety)
Description: as for outcome 12
Time Frame: Participants will be followed for the duration of ICU stay, an expected average of 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 13 | 1

14. Secondary Outcome: Participants With Any Hypoglycemia (<60 mg/dL), Unrelated to Insulin Infusion (Insulin Algorithm Safety)
Description: as for outcome 12
Time Frame: Participants will be followed for the duration of ICU stay, an expected average of 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 26 | 29

15. Secondary Outcome: Participants With Any Hypoglycemia (<60 mg/dL), Related to Insulin Infusion (Insulin Algorithm Safety)
Description: as for outcome 12
Time Frame: Participants will be followed for the duration of ICU stay, an expected average of 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 64 | 5

16. Secondary Outcome: Participants With Hypokalemia (<2.5 mmol/L)
Description: as for outcome 12
Time Frame: Participants will be followed for the duration of ICU stay, an expected average of 8 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Participants | 76 | 64

17. Secondary Outcome: Nursing Workload: SWAT (Subjective Workload Assessment Technique) Instrument
Description: The workload burden placed upon bedside nurses when managing a patient on TGC will be described. Bedside nurses will be randomly selected to complete an anonymous survey describing their perceptions of workload burden associated with managing a patient during one shift.
  Using the SWAT (Subjective Workload Assessment Technique) instrument, perceived workload of Pediatric Intensive Care Nurses caring for HALF-PINT patients in TGC group 1 and TGC group 2 were assessed. The SWAT has been used to study the effect of workload in the fields of nursing, pharmacy and medicine. It measures the following burdens: cognitive (mental effort or concentration required for complexity of task), time (amount of spare time, interruptions, overlapping tasks) and psychological stress associated with work that impacts performance. The SWAT uses a ranking system to weight perceived workload which results in an overall score ranging from 0-100, where higher scores indicate higher perceived workload.
Time Frame: One nursing shift caring for patient on TGC, at anytime during the patient's hospital stay through the tenth nursing shift for the patient. Shift determined randomly by the last digit of the study ID number, 0-9 (0=shift 10, 1=shift 1, 2=shift 2, etc.).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Perceived Nursing Workload: Caring for TGC Group 1 Patients: Approximately half of the subjects randomized into HALF-PINT will be randomized into TGC-1 which will seek to maintain the subject's blood sugar between 80-110 mg/dL. Intravenous insulin may be administered per insulin algorithm. The nurses surveyed were caring for a patient in this treatment arm.
- Perceived Nursing Workload: Caring for TGC Group 2 Patients: Approximately half of the subjects randomized into HALF-PINT will be randomized into TGC-2 which will seek to maintain the subject's blood sugar between 150-180 mg/dL. Intravenous insulin may be administered per insulin algorithm. The nurses surveyed were caring for a patient in this treatment arm.
Arm/Group | Perceived Nursing Workload: Caring for TGC Group 1 Patients | Perceived Nursing Workload: Caring for TGC Group 2 Patients
Number analyzed (Participants) | 250 | 255
score on a scale | 50.0 [24.36 to 60.5] | 36.2 [10.5 to 50.0]

18. Secondary Outcome: Nursing Workload: NASA-TLX (National Aeronautics and Space Administration - Task Load Index) Instrument
Description: The cognitive burden placed upon bedside nurses when managing a patient on TGC will be described. Bedside nurses will be randomly selected to complete an anonymous survey describing their perceptions of workload burden associated with managing a patient on TGC.
  Using the NASA-TLX instrument, perceived workload of Pediatric Intensive Care Nurses caring for HALF-PINT patients in TGC group 1 and TGC group 2 were assessed. The instrument uses a ranking system to weight perceived workload which results in an overall sore ranging from 0-100, where higher scores indicate higher perceived workload. It obtains overall perception of workload related to stressful tasks and includes 6 dimensions (cognitive demand, physical demand, time pressure, performance, effort, and frustration.
Time Frame: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Perceived Nursing Workload: Caring for TGC Group 1 Patients | Perceived Nursing Workload: Caring for TGC Group 2 Patients
Number analyzed (Participants) | 250 | 255
score on a scale | 35.0 [15.3 to 50.0] | 20.4 [7.3 to 38.2]

19. Secondary Outcome: Insulin Algorithm Performance: Time to the Target Range
Description: Performance of the algorithm across diverse ages, weights and disease processes will be critical to measure and compare to other published algorithm performance. Ideally, the algorithm will minimize time to glucose target range. We will track the overall glycemic profile using time-weighted glucose average because it is uniquely unaffected by the increased frequency of BG determinations that occur when glucose is abnormally low or high.
Time Frame: Until study discharge, up to 28 days following randomization
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Hours | 5.5 [2.5 to 11.5] | 1.5 [0.5 to 3.0]

20. Secondary Outcome: Insulin Algorithm Performance: Time in the Target Range
Description: Performance of the algorithm across diverse ages, weights and disease processes will be critical to measure and compare to other published algorithm performance. Ideally, the algorithm will maximize time spent in the glucose target range. We will track the overall glycemic profile using time-weighted glucose average because it is uniquely unaffected by the increased frequency of BG determinations that occur when glucose is abnormally low or high.
Time Frame: Until study discharge, up to 28 days following randomization
Measure: Median (Inter-Quartile Range); unit: Percentage of time
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
Percentage of time | 57 [43 to 67] | 91 [81 to 96]

21. Secondary Outcome: Insulin Algorithm Performance: Time-Weighted Glucose Average
Description: Performance of the algorithm across diverse ages, weights and disease processes will be critical to measure and compare to other published algorithm performance. We will track the overall glycemic profile using time-weighted glucose average because it is uniquely unaffected by the increased frequency of BG determinations that occur when glucose is abnormally low or high.
Time Frame: Until study discharge, up to 28 days following randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Number analyzed (Participants) | 349 | 349
mg/dL | 109 [102 to 118] | 123 [108 to 142]

ADVERSE EVENTS:
Time Frame: Entire course of protocol, up to 28 days
Arm/Group | Tight Glycemic Control 1 (TGC-1) | Tight Glycemic Control 2 (TGC-2)
Serious Adverse Events (participants affected / at risk) | 18/349 | 7/349
Other Adverse Events (participants affected / at risk) | 122/349 | 112/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tight Glycemic Control 1 (TGC-1) (N=349) | Tight Glycemic Control 2 (TGC-2) (N=349)
Severe hypoglycemia (BG < 40 mg/dL) Unrelated to insulin administration (Endocrine disorders) | 5 | 6
Severe hypoglycemia (BG < 40 mg/dL) Related to insulin administration (Endocrine disorders) | 13 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tight Glycemic Control 1 (TGC-1) (N=349) | Tight Glycemic Control 2 (TGC-2) (N=349)
Hypokalemia (< 2.5 mmol/L) (Endocrine disorders) | 76 | 64
New seizure (Nervous system disorders) | 5 | 10
Health-care associated infection (Infections and infestations) | 12 | 4
Infection with positive culture (Infections and infestations) | 29 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No